CLINICAL TRIAL: NCT03382600
Title: A Phase IIb, Clinical Trial to Study the Safety and Efficacy of Pembrolizumab (MK-3475) in Combination With TS-1+Cisplatin or TS-1+Oxaliplatin as a First Line Chemotherapy in Participants With Advanced or Recurrent Gastric Cancer (KEYNOTE-659)
Brief Title: Safety and Efficacy of Pembrolizumab (MK-3475) in Combination With TS-1+Cisplatin or TS-1+Oxaliplatin as First Line Chemotherapy in Gastric Cancer (MK-3475-659/KEYNOTE-659)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3475-659; MK-3475-659 (Other: Merck); KEYNOTE-659 (Other: Merck)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Oxaliplatin; titanium silicide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) (Experimental): Participants receive pembrolizumab 200 mg every 3 weeks (Q3W) plus oxaliplatin 130 mg/m^2 Q3W by intravenous (IV) infusion plus TS-1 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days. Study treatment will be started on Day 1 of each 3-week course, and will continue for up to ~3 years.
  Interventions: Biological: Pembrolizumab; Drug: Oxaliplatin; Drug: TS-1
- Pembrolizumab + Cisplatin +TS-1 (Cohort 2) (Experimental): Participants receive pembrolizumab 200 mg Q3W plus cisplatin 60 mg/m^2 Q3W by IV infusion plus TS-1 BID by continuous oral administration for 14 days, followed by a recovery period of 7 days. Study treatment will be started on Day 1 of each 3-week course, and will continue for up to ~3 years.
  Interventions: Biological: Pembrolizumab; Drug: TS-1; Drug: Cisplatin

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg Q3W on Day 1 by IV infusion
  Other Names: MK-3475
Drug: Oxaliplatin — 130 mg/m^2 Q3W on Day 1 by IV infusion
  Arms: Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1)
Drug: TS-1 — 40 to 60 mg orally according to Body Surface Area (BSA) BID Q3W on Days 1-14
Drug: Cisplatin — 60 mg/m^2 Q3W on Day 1 by IV infusion
  Arms: Pembrolizumab + Cisplatin +TS-1 (Cohort 2)

SUMMARY:
The purpose of this study is to estimate objective response rates (ORRs) of pembrolizumab + oxaliplatin + TS-1 and pembrolizumab + cisplatin + TS-1, as first-line treatment for gastric cancer in programmed death-ligand 1 (PD-L1) positive, human epidermal growth factor receptor 2 (HER2/neu)-negative participants with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
Approximately 45 participants will be assigned to pembrolizumab + oxaliplatin + TS-1 combination therapy (Cohort 1) first, and then 45 participants will be assigned to pembrolizumab + cisplatin + TS-1 combination therapy (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma
* Has a PD-L1 positive tumor as determined by immunohistochemistry (IHC) at a central laboratory
* Has measurable disease as defined by RECIST 1.1 as determined by investigator assessment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at the timing of enrollment
* Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
* Has adequate organ function

Exclusion Criteria:

* Has squamous cell or undifferentiated gastric cancer
* HER2-positive status
* Has had previous therapy for locally advanced, unresectable or metastatic gastric/GEJ cancer
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation
* Has received prior therapy with a platinum-based anti-cancer drug
* Has had major surgery, open biopsy or significant traumatic injury within 28 days prior to enrollment, or anticipation of the need for major surgery during the course of study treatment
* Has had radiotherapy within 14 days of enrollment
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years with use of disease modifying agents, corticosteroids, or immunosuppressive drugs
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has any active infection requiring systemic therapy
* Will be on flucytosine at the time of enrollment
* Has grade ≥ 2 peripheral sensory neuropathy
* Has poorly controlled diarrhea (e.g., watery stool, uncontrollable bowel movement with drugs, grade ≥ 2 and number of defecations, ≥ 5/day)
* Has accumulation of pleural, ascitic, or pericardial fluid requiring drainage within 2 weeks prior to enrollment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has known history of human immunodeficiency virus (HIV) [HIV1/2 antibodies]
* Has a known history of Hepatitis B
* Has received live vaccine within 30 days of the planned start of study therapy
* Is currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of trial treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- Japan (25):
  - National Cancer Center Hospital East ( Site 0001), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0024), Matsuyama, Ehime
  - Gunma Prefectural Cancer Center ( Site 0005), Ohta, Gunma
  - Hokkaido University Hospital ( Site 0006), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 0016), Akashi, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 0015), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 0018), Kasama, Ibaraki
  - Kitasato University Hospital ( Site 0019), Sagamihara, Kanagawa
  - Kanagawa Cancer Center ( Site 0003), Yokohama, Kanagawa
  - Tohoku University Hospital ( Site 0023), Sendai, Miyagi
  - Kindai University Hospital ( Site 0013), Sayama, Osaka
  - Osaka University Hospital ( Site 0010), Suita, Osaka
  - Saitama Cancer Center ( Site 0004), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0020), Sunto-gun, Shizuoka
  - Jichi Medical University Hospital ( Site 0009), Shimotsuke, Tochigi
  - Chiba Cancer Center ( Site 0012), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0017), Fukuoka
  - Kyushu University Hospital ( Site 0014), Fukuoka
  - Gifu University Hospital ( Site 0021), Gifu
  - Kochi Health Sciences Center ( Site 0022), Kochi
  - Kumamoto University Hospital ( Site 0002), Kumamoto
  - Osaka International Cancer Institute ( Site 0011), Osaka
  - National Cancer Center Hospital ( Site 0025), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0008), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0007), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] https://pubmed.ncbi.nlm.nih.gov/35701865/
- [Derived] Kawazoe A, Yamaguchi K, Yasui H, Negoro Y, Azuma M, Amagai K, Hara H, Baba H, Tsuda M, Hosaka H, Kawakami H, Oshima T, Omuro Y, Machida N, Esaki T, Yoshida K, Nishina T, Komatsu Y, Han SR, Shiratori S, Shitara K. Safety and efficacy of pembrolizumab in combination with S-1 plus oxaliplatin as a first-line treatment in patients with advanced gastric/gastroesophageal junction cancer: Cohort 1 data from the KEYNOTE-659 phase IIb study. Eur J Cancer. 2020 Apr;129:97-106. doi: 10.1016/j.ejca.2020.02.002. Epub 2020 Mar 4. PMID 32145474
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Programmed cell death ligand 1 (PD-L1) positive, human epidermal growth factor receptor 2 (HER2)/neu negative participants 18 to 75 years of age with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma were recruited at 25 study sites in Japan.
Groups:
- Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1): Participants received pembrolizumab 200 mg every 3 weeks (Q3W) plus oxaliplatin 130 mg/m^2 Q3W by intravenous (IV) infusion plus TS-1 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days. Study treatment started on Day 1 of each 3-week course, and continued for up to ~3 years.
- Pembrolizumab + Cisplatin +TS-1 (Cohort 2): Participants received pembrolizumab 200 mg Q3W plus cisplatin 60 mg/m^2 Q3W by IV infusion plus TS-1 BID by continuous oral administration for 14 days, followed by a recovery period of 7 days. Study treatment started on Day 1 of each 3-week course, and continued for up to ~3 years.
Period: Overall Study
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Started | 54 | 46
Completed | 0 | 0
Not Completed | 54 | 46
Not completed — Adverse Event | 3 | 3
Not completed — Clinical Disease Progression | 2 | 4
Not completed — Radiological Progression | 40 | 31
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1): Participants received pembrolizumab 200 mg Q3W plus oxaliplatin 130 mg/m^2 Q3W by IV infusion plus TS-1 BID by continuous oral administration for 14 days, followed by a recovery period of 7 days. Study treatment started on Day 1 of each 3-week course, and continued for up to ~3 years.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2) | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.6) | 62.9 (10.2) | 62.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 43 | 28 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 54 | 46 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR)
Description: For the primary efficacy analysis, ORR was defined as the percentage of participants who have a best response of complete response (CR, disappearance of all target lesions) or partial response (PR, at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) per RECIST 1.1 as assessed by BICR.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Percentage of participants | 72.2 [58.4 to 83.5] | 80.4 [66.1 to 90.6]

2. Secondary Outcome: ORR According to Immune-related Response Evaluation Criteria In Solid Tumors (iRECIST) Assessed by BICR
Description: For the secondary efficacy analysis, ORR was defined as the percentage of participants whose best response based on imaging is CR (disappearance of all target lesions) or PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to iRECIST as assessed by BICR. iRECIST is a modification to RECIST that takes into account unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Percentage of participants | 72.2 [58.4 to 83.5] | 80.4 [66.1 to 90.6]

3. Secondary Outcome: Duration of Response (DOR) According to RECIST 1.1 Assessed by BICR
Description: For participants who demonstrated complete response (CR, disappearance of all target lesions) or partial response (PR, ≥30% decrease in the SOD of target lesions) according to RECIST 1.1 as assessed by BICR, DOR was defined as the time from the earliest date of qualifying response (CR or PR) until earliest date of progressive disease (PD, ≥20% increase in the SOD of target lesions) or death from any cause, whichever came first. DOR was censored at the last tumor assessment date if a responder did not have PD or death.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug and had a confirmed response of CR or PR are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 39 | 37
months | 10.6 [5.6 to NA] — Insufficient events to calculate the upper bound of the confidence interval. | 9.5 [4.7 to 15.3]

4. Secondary Outcome: DOR According to iRECIST Assessed by BICR
Description: For participants who demonstrated complete response (CR, disappearance of all target lesions) or partial response (PR, ≥30% decrease in the SOD of target lesions) according to iRECIST as assessed by BICR, DOR was defined as the time from the earliest date of qualifying response (CR or PR) until earliest date of progressive disease (PD, ≥20% increase in the SOD of target lesions) or death from any cause, whichever came first. DOR was censored at the last tumor assessment date if a responder did not have PD or death. iRECIST is a modification to RECIST that takes into account unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug and had a confirmed response of CR or PR are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 39 | 37
months | 10.6 [5.6 to NA] — Insufficient events to calculate the upper bound of the confidence interval. | 9.5 [4.7 to NA] — Insufficient events to calculate the upper bound of the confidence interval.

5. Secondary Outcome: Disease Control Rate (DCR) According to RECIST 1.1 Assessed by BICR
Description: DCR was defined as the percentage of participants in the analysis population who have complete response (CR, disappearance of all target lesions), partial response (PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline SOD), or stable disease (SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD, ≥20% increase in the SOD of target lesions]). Responses are according to RECIST 1.1 as assessed by BICR.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Percentage of participants | 96.3 [87.3 to 99.5] | 97.8 [88.5 to 99.9]

6. Secondary Outcome: DCR According to iRECIST 1.1 Assessed by BICR
Description: DCR was defined as the percentage of participants in the analysis population who have CR (disappearance of all target lesions), PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline SOD), or stable disease (SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [≥20% increase in the SOD of target lesions]). Responses are according to iRECIST 1.1 as assessed by BICR. iRECIST is a modification to RECIST that takes into account unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Percentage of participants | 96.3 [87.3 to 99.5] | 97.8 [88.5 to 99.9]

7. Secondary Outcome: Time to Response (TTR) According to RECIST 1.1 Assessed by BICR
Description: TTR was defined as the time from the date of enrollment day to the first date of confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline SOD). Responses are according to RECIST 1.1 as assessed by BICR.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
months | 1.5 [1.3 to 5.5] | 1.5 [1.2 to 2.9]

8. Secondary Outcome: TTR According to iRECIST 1.1 Assessed by BICR
Description: TTR was defined as the time from the date of enrollment day to the first date of confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline SOD). Responses are according to iRECIST 1.1 as assessed by BICR. iRECIST is a modification to RECIST that takes into account unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
months | 1.5 [1.3 to 5.5] | 1.5 [1.2 to 2.9]

9. Secondary Outcome: Progression-free Survival (PFS) According to RECIST 1.1 Assessed by BICR
Description: PFS was defined as the time from the date of enrollment day to the first documented PD (defined as ≥20% increase in the SOD of target lesions) or death due to any cause, whichever occurred first. Responses are according to RECIST 1.1 as assessed by BICR.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
months | 9.4 [6.6 to 12.6] | 8.3 [5.8 to 15.3]

10. Secondary Outcome: PFS According to iRECIST 1.1 Assessed by BICR
Description: PFS was defined as the time from the date of enrollment day to the first documented PD (defined as ≥20% increase in the SOD of target lesions) or death due to any cause, whichever occurred first. Responses are according to iRECIST 1.1 as assessed by BICR. iRECIST is a modification to RECIST that takes into account unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
months | 9.4 [6.6 to 12.6] | 10.9 [6.7 to NA] — Insufficient events to calculate the upper bound of the confidence interval.

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of enrollment day to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. For these participants, date of last follow up was last visit date instead of death date.
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
months | 16.9 [13.4 to 20.0] | 17.1 [12.6 to 23.1]

12. Secondary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Participants | 54 | 46

13. Secondary Outcome: Number of Participants Discontinuing From Study Treatment Due to AE(s)
Description: as for outcome 12
Time Frame: Up to ~36 months
Population: All participants who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
Number analyzed (Participants) | 54 | 46
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to ~36 months
Description: All participants who received ≥1 dose of study drug are included. Per protocol, disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", "Disease progression" unrelated to study drug are excluded as AEs.
Arm/Group | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 3/54 | 0/46
Serious Adverse Events (participants affected / at risk) | 27/54 | 22/46
Other Adverse Events (participants affected / at risk) | 54/54 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) (N=54) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2) (N=46)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cytomegalovirus enterocolitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Oxaliplatin +TS-1 (Cohort 1) (N=54) | Pembrolizumab + Cisplatin +TS-1 (Cohort 2) (N=46)
Anaemia (Blood and lymphatic system disorders) | 13 | 18
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 6
Vertigo (Ear and labyrinth disorders) | 3 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 3
Hypothyroidism (Endocrine disorders) | 5 | 3
Cataract (Eye disorders) | 0 | 3
Lacrimation increased (Eye disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 4
Colitis (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 24 | 30
Diarrhoea (Gastrointestinal disorders) | 24 | 22
Nausea (Gastrointestinal disorders) | 34 | 28
Stomatitis (Gastrointestinal disorders) | 16 | 17
Vomiting (Gastrointestinal disorders) | 13 | 11
Fatigue (General disorders) | 12 | 15
Malaise (General disorders) | 22 | 15
Oedema (General disorders) | 5 | 4
Oedema peripheral (General disorders) | 8 | 7
Pyrexia (General disorders) | 13 | 10
Infusion site extravasation (General disorders) | 0 | 3
Hypersensitivity (Immune system disorders) | 3 | 0
Bronchitis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 8
Pneumonia (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 9 | 6
Aspartate aminotransferase increased (Investigations) | 12 | 9
Blood bilirubin increased (Investigations) | 4 | 2
Blood creatinine increased (Investigations) | 1 | 6
Gamma-glutamyltransferase increased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 24 | 32
Platelet count decreased (Investigations) | 29 | 11
Weight decreased (Investigations) | 7 | 5
Weight increased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 8 | 10
Blood alkaline phosphatase increased (Investigations) | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 7
Decreased appetite (Metabolism and nutrition disorders) | 38 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 5
Dysgeusia (Nervous system disorders) | 19 | 15
Headache (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 51 | 14
Insomnia (Psychiatric disorders) | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 10
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 6
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Embolism (Vascular disorders) | 2 | 3
Vascular pain (Vascular disorders) | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03382600/Prot_SAP_000.pdf